# **Protocol**

**Study ID:** 213550

**Official Title of Study:** COPD disease burden, patient characteristics, maintenance treatment patterns and factors influencing treatment decisions in China Tier 2 and Tier 3 hospitals

**NCT ID:** NCT04853238

**Date of Document:** 26-May-2022

## CONFIDENTIAL



# **HEALTH OUTCOMES STUDY PROTOCOL - QUALITATIVE RESEARCH**

| UNIQUE IDENTIFIER | 213550 |
|---|---|
| FULL TITLE | COPD disease burden, patient characteristics, maintenance |
| | treatment patterns and factors influencing treatment |
| | decisions in China Tier 2 and Tier 3 hospitals |
| ABBREVIATED TITLE | COPD maintenance treatment patterns in China |
| FINAL PROTOCOL APPROVED | |
| SPONSORSHIP | Sponsored |
| DIVISION | Pharma |
| BUSINESS UNIT | Medical Affairs |
| DEPARTMENT | Medical Affairs |
| STUDY ACCOUNTABLE PERSON | PPD |
| CONTRIBUTING AUTHORS | |

| ASSET ID | GSK2834425, GW685698/GW642444/GSK573719 |
|------------|-----------------------------------------|
| GSK ASSET | Trelegy |
| INDICATION | Chronic Obstructive Pulmonary Disease |

# **REVISION CHRONOLOGY:**

| Version Date Docu | ment Type | Change(s) since last version |
|-------------------|------------|------------------------------|
| Versi | on ID: 2.0 | 1.0 |

Description: COPD maintenance treatment patterns in China

Unique Identifier: 213550

# **SPONSOR SIGNATORY**

| PPD | |
|----------------------------------------------|------|
| [Xiao Hu], Medical Affairs Manager | Date |
| Primary Author/ Project officer | |
| PPD | |
| [Jody Goh], Head of Respiratory Therapy Area | Date |
| PPD | |
| [ Pauling Ng], Country Medical Director | Date |

Description: COPD maintenance treatment patterns in China

Unique Identifier: 213550

# **Investigator Protocol Agreement Page**

- I confirm agreement to conduct the study in compliance with the protocol.
- I acknowledge that I am responsible for overall study conduct. I agree to personally conduct or supervise the described clinical study.
- I agree to ensure that all associates, colleagues and employees assisting in the conduct of the study are informed about their obligations. Mechanisms are in place to ensure that site staff receives the appropriate information throughout the study.

| Investigator Name: | |
|------------------------|--------------------|
| <del></del> | |
| Investigator Signature | Date (DD-MMM-YYYY) |

# **PROTOCOL SYNOPSIS**

| Unique Identifier | 213550 |
|---|---|
| Abbreviated Title | COPD maintenance treatment patterns in China |
| GSK Product | Trelegy |
| Rationale | Pharmacological treatment of COPD, as perceived by physicians in China, appears very complicated, especially with the increasing number of therapeutic options available and recommendations to personalise treatment of COPD patients to individual needs. Physicians also use different treatment strategies for symptom reduction and exacerbation prevention. For example, many use a step-up approach but some use intensive treatment initially, followed by step down. In addition, treatments depend on the socioeconomic condition of the patient such as occupation, educational level, income and environment. |
| | A further complication in China is that there are different tiers of hospitals with different formularies and patients move between hospitals and doctors very readily. In addition, the re-attendance rate to the same clinic/physician is low, resulting in little continuity of care. Therefore, this study is conducted to gain an adequate understanding of the complex COPD management environment and |
| Objectives | doctors' treatment strategy of COPD in China. Primary |
| (Primary, Secondary) | To quantify the pattern of COPD maintenance treatment prescribing in different patient groups in Tier 2 and 3 hospitals in China Secondary To examine factors (including disease severity and socio- |
| | <ul> <li>economic factors) that are associated with different patterns of COPD maintenance treatment</li> <li>To assess the proportion of patients whose prescribed maintenance treatment is stepped up, stepped down, switched, stopped or remains the same across the different study time points</li> <li>Assess the disease burden of the patients</li> </ul> |

| <ul> <li>To assess the proportion of patients receiving each treatment<br/>class at 3 months.</li> </ul> |
|---|
| This will be a 3-month, multicentre, prospective, low-interventional |
| study in newly diagnosed and previously diagnosed patients with |
| COPD presenting to clinics, either in stable state or with an acute |
| exacerbation, in Tier 2 and 3 hospitals in China. The study will be |
| conducted at around 35 sites (±5 sites). For the primary analysis, |
| the patients will be categorised into 3 cohorts: |
| 1. Cohort 1: Patients presenting with stable disease |
| 2. Cohort 2: Patients presenting with a moderate exacerbation |
| not requiring hospitalization |
| 3. Cohort 3: Patients requiring hospitalisation for an |
| exacerbation |
| Inclusion Criteria |
| Male or female patients with ≥40 years of age at the time of signing |
| the informed consent with a diagnosis of COPD confirmed by |
| spirometry (According to GOLD 2019 criteria). |
| Exclusion Criteria |
| Patients with a current primary diagnosis of asthma, active |
| tuberculosis, bronchiectasis, lung cancer or other active |
| pulmonary disease, other unstable diseases or cognitive |
| behaviour, which could influence COPD assessment test |
| (CAT) and lung function results in the view of their |
| physicians. |
| Patients who experienced a physician-treated moderate or |
| severe COPD exacerbation within the last 1 month before |
| screening. |
| Patient participating in another COPD clinical study using |
| investigational medication and/or disease management |
| process. |
| Primary Endpoints |
| The data source will be the study case record form (CRF) |
| COPD prescription for maintenance therapy (Long-Acting |
| Muscarinic Antagonist [LAMA], Long-Acting Beta-Agonist |
| [LABA]; dual bronchodilator, inhaled corticosteroid [ICS]/ Long- |
| Acting Beta-Agonist [LABA], triple therapy, theophylline and n- |

• COPD prescription for maintenance therapy collected at 3 months (all patients) and at 1 week after a moderate exacerbation or on discharge following hospitalisation.

## **Secondary Endpoints**

- Data source mentioned in primary endpoints
- FEV1, exacerbations in previous 1 year, CAT score, Modified Medical Research Council (mMRC) score, co-morbidity, socioeconomic status, COPD medication history (within past 1 month)

## Data Analysis Methods

The number and percentage of patients who use the maintenance treatment at each visit will be summarized. Moreover, for those who use maintenance treatment, the number and percentage of patients will be summarized for each of the following pattern of maintenance treatment:

- Long-Acting Muscarinic Antagonist [LAMA]
- Long-Acting Beta-Agonist [LABA]
- Dual bronchodilator
- Inhaled corticosteroid [ICS]/ Long-Acting Beta-Agonist [LABA]
- Triple therapy
- Theophylline
- N-acetyl cysteine/carbocysteine

The results for patients with stable disease and patients with exacerbation at baseline will be analysed separately for the following visits: baseline visit, 1-week follow up (for moderate exacerbations) and discharge follow-up (for hospitalised exacerbations). The results for patients with stable disease and patients with exacerbation will be pooled together for analysis for 3-month follow-up visit.

#### Sample Size and Power

For this study, around 1500 patients with COPD will be enrolled including stable patients (~50% of the total patients) and patients with exacerbations (~50% of the total patients). All enrolled patients will be included in the analysis. A large overall sample size was chosen to ensure adequate patient representation across China. It is estimated that 750 patients each from tier 2 and tier 3 hospitals will be enrolled to provide adequate representation on healthcare status for COPD in China. After 500 patients have been

| recruited, the numbers will be reviewed to assess whether an |
|---------------------------------------------------------------------|
| adequate number of patients from each of the 3 cohorts have been |
| enrolled for each tier of hospital. Recruitment policy might be |
| changed to ensure an adequate distribution of patients. |
| Potential limitations have been listed below. |
| 1) The study has covered major Chinese provinces as |
| comprehensively as possible, choosed 1-2 sites from major |
| Chinese province but this may not be fully representative of all |
| the Tier 2&3 hospitals in each province. |
| 2) The study includes only those Tier 2 hospitals at a minimum |
| have respiratory department which have LAMA and ICS/LABA |
| and spirometry available; however, this will not fully reflect |
| COPD management in all Tier 2 hospitals, because not all |
| currently have such drugs available. This situation is changing so |
| that all Tier 2 hospitals will have these treatments available |
| relatively soon. |
| 3) It is a 3-month follow-up study and the duration is adequate to |
| measure short-medium term changes, but COPD requires |
| lifelong treatment, so this reflects only a short period of a |
| patient's management. |
| 4) The adherence data is reliant on the patients accurate reporting |
| of which prescribed treatments they are taking, there can be an |
| underestimation or overestimation of adherence to medication. |

## **TABLE OF CONTENTS**

| PROTOCOL SYNOPSIS | 4 |
|--------------------------------------------------------------------|----|
| TABLE OF CONTENTS | 8 |
| ABBREVIATIONS | 9 |
| 1 INTRODUCTION/BACKGROUND | 12 |
| 2 RESEARCH OBJECTIVES | 14 |
| 2.1 Primary Objective: | 14 |
| 2.2 Secondary Objectives | 14 |
| CCI | |
| 3 RESEARCH METHODOLOGY | 15 |
| 3.1 Study Design | 15 |
| 3.2 Study Population | 16 |
| 3.2.1 Eligibility Criteria | 16 |
| 3.2.2 Sampling | 17 |
| 3.3 Data Source / Data Collection | |
| 3.3.1 Endpoints data source | 22 |
| 3.3.2 Exposure and outcomes | 23 |
| 4 SAMPLE SIZE / POWER CALCULATIONS | 27 |
| 4.1 Hypotheses | 28 |
| 5 DATA ANALYSIS CONSIDERATIONS | 28 |
| 5.1 Primary analyses | 28 |
| 5.2 Secondary analyses | 29 |
| CCI | |
| 5.4 Other analysis | |
| 6 LIMITATIONS | |
| 7 STUDY CONDUCT, MANAGEMENT & ETHICS | 31 |
| 7.1 Ethics Committee/IRB Approval | 31 |
| 7.2 Informed Consent | |
| 7.3 Data Protection | |
| 7.4 Personally Identifiable Information (PII) | 32 |
| 7.5 Adverse Event (AE), Pregnancy Exposure, and Incident Reporting | |
| 7.6 Legal Basis for Processing Individual Human Data | |
| 8 PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | 33 |
| 8.1 Target Audience | 33 |
| 8.2 Study reporting and publications | |
| 9 REFERENCES | |
| 10 APPENDICES | |
| 10.1 Appendix 1: SCHEDULE OF ACTIVITIES | 36 |

| Appendix 2: COPD assessment test | 40 |
|---|---|
| Appendix 3: Modified British Medical Research Council (mMRC) Dyspnoea Scale | 42 |
| Appendix 4: DECAF score | 43 |
| Appendix 5: Patient survey and questionnaire | 44 |
| Economics Information: | 44 |
| Knowledge: | 45 |
| on't go for follow-up visits regularly, why not? (Choose as many as you want) | 46 |
| ns (PHQ9): | 48 |
| Economics Information: | 50 |
| Knowledge: | 50 |
| ns (PHQ9):: | 53 |
| Appendix 6: sPVP and PVP APPROVAL FORM | 55 |
| | Appendix 3: Modified British Medical Research Council (mMRC) Dyspnoea Scale |

# **ABBREVIATIONS**

| AE | Adverse Event |
|-------------|------------------------------------------------------------|
| BMI | Body Mass Index |
| CAT | COPD assessment test |
| CE | Concept Elicitation |
| CFR | Code of Federal Regulations |
| CI | Confidence Interval |
| COPD | Chronic Obstructive Pulmonary Disease |
| CRF | Case Report Form |
| CVD | Cardiovascular Disease |
| DECAF Score | Dyspnoea, Eosinopenia, Consolidation, Acidaemia and atrial |
| | Fibrillation (DECAF) Score |
| eMRCD | Extended MRC Dyspnea Scale |
| ER | Emergency room |
| FEV1 | Forced expiratory volume in one minute |
| FSFV | First subject first visit |
| GCP | Good Clinical Practice |
| GERD | Gastroesophageal Reflux Disease |
| GSE | General Self-Efficacy Scale |
| GP | General Physician |
| GSK | GlaxoSmithKline |
| HIPAA | Health Insurance Portability and Accountability Act |
| ICF | Informed Consent Form |

| ICH | International Conference on Harmonization |
|------|-----------------------------------------------|
| ICS | Inhaled corticosteroid |
| IEC | Independent Ethics Committee |
| IHD | Individual human data |
| IPAQ | International physical activity questionnaire |
| IRB | Institutional Review Board |
| LABA | Long-acting beta agonists |
| LAMA | Long-acting muscarinic antagonist |
| LSLV | Last subject's last visit |
| mMRC | Modified Medical Research Council |
| OR | Odds Ratio |
| OSAS | Obstructive Sleep Apnea Syndrome |
| SAMA | Short-acting muscarinic antagonist |
| SABD | Short acting bronchodilator |
| OPD | Outpatient department |
| PHQ9 | The patient health questionnaire |
| PI | Principle Investigator |
| PII | Personally Identifiable Information |
| PRO | Patient Reported Outcome |
| PVP | Pharmacovigilance Program |
| V | Visit |

# **Trademark Information**

# Trademarks of the GlaxoSmithKline group of companies

COPD assessment test (CAT)

Trademarks not owned by the GlaxoSmithKline group of companies

## 1 INTRODUCTION/BACKGROUND

Chronic obstructive pulmonary disease (COPD) is a preventable and treatable disease characterized by persistent respiratory symptoms and airflow limitation that is due to airway and/or alveolar abnormalities usually caused by significant exposure to noxious particles or gases [GOLD, 2019]. This is associated with increased morbidity and risk of early death [Agusti, 2005; Qaseem, 2011; Rodríguez, 2010].

COPD is the third most prevalent disease in China after hypertension and diabetes [Wang 2018]. A study conducted between 2012-2015 found that 8.6% of Chinese aged ≥20 years met spirometry-defined COPD criteria and the COPD prevalence in adults ≥40 years was 13.7%. This amounts to 99.9 million people with potential COPD in China [Wang, 2018]. Annually, around 8 million Chinese patients are hospitalised due to COPD exacerbations, but a larger but unquantified number of patients experiencing moderate exacerbations are treated as an outpatient. A survey in China, reported that the average exacerbation rate in patients diagnosed with COPD was approximately 2.5 exacerbations per year per patient [Jia, 2018]. The frequency of exacerbations may be influenced by patients' level of education and treatment adherence, physicians' treatment decisions and disparity in prescription practice [Cai, 2015; Fang, 2012; Zha, 2019]. The failure of patients and physicians to recognise the significance of exacerbations adds to the challenges in COPD treatment.

Hospitalisation due to COPD exacerbations is associated with high healthcare costs. In China, patients with an acute exacerbation of COPD are admitted to a Tier-3 hospital with an average total cost of \$1323 per admission [Yang, 2012]. Reducing hospitalisation through more effective maintenance treatment would greatly reduce healthcare costs in China. Appropriate management of COPD starts with diagnosis. In a study conducted in Beijing, 29% of the patients with high-risk COPD were undiagnosed [Rui, 2014] and many physicians do not consider spirometry as the most appropriate test when a diagnosis of COPD is suspected [Wang, 2018].

In China, there are three tiers of hospital. Tier 1 hospitals have very basic facilities and limited formularies for the long-term management of COPD. Tier 2 hospitals have more facilities and get access to a wider range of treatments, which usually includes the main treatment classes for COPD, but not the latest therapies. The Tier 3 hospitals have the full range of COPD therapies; however, the government is actively encouraging a shift of COPD patients from Tier 3 to Tier 2 hospitals. One more complication in China is that patients move between hospitals and doctors very readily, resulting in very little continuity of care. The experts with an interest in COPD are in a view that the re-attendance rate to the same clinic/physician is very low (approx below 50%).

In a prescription survey conducted between 2010 and 2011 in China, it was observed that, as elsewhere in the world, physicians do not follow GOLD recommendations. [Fang, 2012]. In

addition, the economic burden poses a big challenge, since the social insurance bureau and private companies in China generally reimburse treatment costs due to hospitalisation, rather than maintenance treatment. Such policies are one of the leading causes of under-prescribing of drugs by physicians, because patients fail to receive adequate reimbursement [Li, 2018] and this leads to suboptimal treatment.

Another important factor is the patients' adherence to maintenance therapy, which remains a substantial barrier to optimal disease control. Despite evidence that adherence to inhaled COPD therapy is associated with improved symptom control, lung function and reductions in healthcare resource utilisation and costs, patients non-compliance to treatment remains a major problem [Davis, 2017;

Mäkelä, 2013; Toy, 2011]. Studies in patients with COPD in the Western countries have shown that around 50% patients have suboptimal adherence to treatment [Restrepo, 2008], this is likely to be further low in China, due to low educational qualification of the patient attending COPD units.

Smoking is a major risk factor for COPD. In China, in a study by Jiangna et al, around 82% of the patients recruited in tertiary care hospital were current or ex-smokers. However, there are COPD patients who are never-smokers [GOLD, 2020], due to a range of causes including but not limited to, childhood chest illnesses, passive cigarette, biomass fuel exposure and pollution. Therefore, to ensure an adequate representation of treatment for COPD in China, all patients with a clinical diagnosis of COPD, confirmed on spirometry, will be recruited and their smoking history will be recorded.

#### Rationale

In recent years, physicians in China have perceived pharmacological treatment of COPD to be very complicated, especially with the increasing number of therapeutic options available and recommendations to personalise treatment. Physicians also use different treatment strategies. A further complication is that treatment will depend on socio-economic factors such as occupation, educational level, income and patients' preference. Besides, patients move between hospitals and doctors very readily, resulting in very little continuity of care. The experts with an interest in COPD are in view that the re-attendance rate to the same clinic/physician is very low (approx. below 50%).

To improve COPD management in China, it is important to understand current patterns of COPD medication prescription and assess the effect of patient characteristics and other factors on treatment decisions made by physicians. Whilst data on physicians' prescribing practises can be obtained through surveys or market research, this can't capture the impact of the broad range of factors that a physician may take into account when deciding on treatment for an

individual patient, hence answers to paper-based scenarios may not accurately reflect behaviour in routine practice. In China, there are currently no databases that would permit analysis of prescribing to well characterised COPD patient groups. A prospective study of actual prescribing at an individual patient level is required, coupled with an assessment of the patient's clinical severity and socio-economic status. This will allow a detailed analysis of the maintenance treatment used for different patient groups and give an insight into the factors that physicians take into account when deciding on treatment.

There are three main clinical scenarios seen in Chinese hospitals:

- 1. Patients presenting with stable disease
- 2. Patients presenting with a moderate exacerbation
- 3. Patients requiring hospitalisation for an exacerbation

In each scenario, the patients may be treated differently, so it is necessary to determine prescribing practices of the physician in each case and identify factors associated with the prescription. It is also necessary to know how the maintenance treatment of the patients changes over time, and the level of the patient's adherence to their prescriptions, as this thought to be low in China, but has not been measured.

In China clinical practice, some patients may be admitted to hospital with an exacerbation but not because of the severity of the exacerbation (i.e. by the request of the patient). To ensure that patients are only recruited to the study because of the severity of the exacerbation, an inclusion criterion of the requirement for intravenous therapy is needed, since this treatment cannot be administered at home.

#### **2 RESEARCH OBJECTIVES**

#### 2.1 Primary Objective:

• To quantify the pattern of COPD maintenance treatment prescribing in different patient groups in Tier 2 and 3 hospitals in China

## 2.2 Secondary Objectives

- To examine factors (including disease severity and socio-economic factors) that are associated with different patterns of COPD maintenance treatment
- To assess the disease burden of patients (using baseline data)
- To assess the proportion of patients whose prescribed maintenance treatment is stepped up (adding another maintenance treatment), stepped down (withdraw any of the maintenance medication but kept the maintenance treatment), switch (between

LAMA+LABA and ICS/LABA), stopped (stop all maintenance treatment) or remains the same across the different study time points

• To assess the proportion of patients receiving each treatment class at 3 months



#### 3 RESEARCH METHODOLOGY

## 3.1 Study Design

This will be a 3-month, multicentre, prospective study in newly diagnosed and previously diagnosed patients with COPD presenting to clinics, either in a stable state, defined as no exacerbation for at least 1 month, or with acute exacerbation, in Tier 2 and 3 hospitals distributed across China. The study will be conducted at around 35 sites (±5 sites). The patients will be categorised into 3 cohorts:

- 1. Cohort 1: Patients presenting with stable disease (newly and previously diagnosed)
- 2. Cohort 2: Patients presenting with a moderate acute exacerbation not requiring hospitalization
- 3. Cohort 3: Patients requiring hospitalisation for an acute exacerbation



Tel.-Telephone

Figure 1: The study schematic

At site evaluation (conducted to evaluate if the sites can be included in the study), the types of medical insurance covered by the hospital, types of COPD maintenance medication available to be supplied to patients and reimbursement rate for each out-patient and in-patient medication will be collected before patient recruitment.

## 3.2 Study Population

The study population comprises COPD patients in stable status or with acute exacerbation in tier 2 and tier 3 hospitals. Stable status at enrolment is defined as no exacerbation events in the preceding month. An exacerbation of COPD is as an acute worsening of respiratory symptoms that results in additional therapy. Moderate exacerbation is defined as worsening of symptoms for which a patient seeks medical care and is treated by antibiotics and/or systemic corticosteroids /or corticosteroids nebulization, severe exacerbation is defined as patient requires hospitalization or visits the emergency room (ER)

## 3.2.1 Eligibility Criteria

#### 3.2.1.1 Inclusion Criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

- Patients ≥40 years of age
- Male or female
- A diagnosis of COPD confirmed by spirometry (According to GOLD 2019 criteria) in Tier 2 and Tier 3 hospitals
- In hospitalized patients, recruit only patients who receive any intravenous therapy
- A signed and dated written informed consent must be obtained from the patient prior to study participation
- Patients can communicate normally

#### 3.2.1.2 Exclusion Criteria

A subject who meets any of the following criteria will be excluded from participation in this study:

- Current primary diagnosis of asthma, active tuberculosis, bronchiectasis, lung cancer or other active pulmonary disease
- Other unstable diseases or cognitive behaviour, which could influence CAT and lung function results (judged by physicians)
- Experienced a moderate/severe COPD exacerbation treated by a physician within last 1 month

 Currently participating in another COPD clinical study, which provides the patient investigational medication and/or disease management

## 3.2.2 Sampling

For this study, around 1500 patients with COPD will be enrolled including stable patients and patients with exacerbations. It is planned that approximately equal number of patients will be recruited from Tier 2 and Tier 3 hospitals. After 500 patients have been recruited a review will be carried out to assess whether an adequate number of patients from each of the 3 cohorts defined in section 3.1 has been enrolled. At this point, recruitment policy might be changed to ensure an adequate distribution across type of hospital and type of patient. Thereafter, recruitment to each cohort will be monitored weekly and further corrective action will be taken if needed.

At least one site in each of the main provinces of China will be selected. There is a variability of spirometry and inhaled therapy availability across Tier 2 hospitals, although this is improving. As the Government is actively encouraging patients to shift from Tier 3 to Tier 2 hospitals, the study will only include Tier 2 hospitals that, at a minimum have respiratory department, supply of LAMA and ICS/LABA, and facilities for spirometry, since this will be the minimum standard of care for patients with COPD in Tier 2 hospitals in the future.

#### 3.2.2.1 Patients presenting with stable disease

#### Baseline visit (Day 1):

Newly or previously diagnosed patients with stable COPD who attend the clinic will be screened by the study physician. Once eligible patients have been identified, informed consent will be obtained. The physician will then make their treatment decision, before any other study assessments are made.

This visit will be considered as Baseline visit (V1). During the Baseline visit, the following information will be collected:

- 1. Demography
- 2. Time since first COPD diagnosis
- 3. Co-morbidities
- 4. COPD exacerbation history in prior 12 months
- 5. COPD medication history (within past 1 month)
- 6. Concomitant medication
- 7. COPD medication prescribed at baseline visit (including the drugs prescribed this time and the drugs that the subject needs to continue to use)

- 8. Smoking history
- 9. Spirometry (within 7 days of enrollment)†
- 10. Modified Medical Research Council (mMRC) dyspnea scale, CAT
- 11. Socio-Economic status (refer to 3.3.2.10)
- 12. Patient questionnaire and survey ††
- 13. Physician survey ††
- 14. Collect spontaneously AE/SAE reports on GSK products
- 15. Maintenance treatment class availability in hospital internal pharmacy+++
- 16. Prescribing physician's name<sup>†††</sup>.
- $\dagger$  FEV<sub>1</sub> performed within 6 months before the index date will be acceptable. Index date is the date when physician collect data for baseline. A 7-day time window was set between the time when the V1 lung function results were obtained and the day of enrollment to ensure that there was sufficient time to obtain the lung function report results to deal with the interference of the COVID-19 epidemic on the study.
- †† Patient questionnaires include International physical activity questionnaire (IPAQ), The patient health questionnaire (PHQ9), General self-efficacy scale. Patient's survey is developed by the study initiator. The physician's survey is developed by the study initiator.
- ††† Data will not be collected from patient

## 3-month Follow-up visit (Day 90 ± 7):

All patients will be followed-up telephonically after 3 months. Following information will be collected:

- 1. Current COPD medication taken by the patient, including prescription of current treatment and time of prescription, physician and hospital name<sup>#</sup>.
- 2. COPD Clinic revisit times and reason
- 3. Frequency of COPD exacerbation between baseline visit and 3 months follow up
- 4. Reason for the last hospital visit (i.e. routine or exacerbation)
- 5. Identify prescribed treatments that the patients did not take on the day of the call\*.
- 6. CAT
- 7. Patient questionnaire and survey †
- 8. Collect spontaneously AE/SAE reports on GSK products

# A photo of the physician's prescription which includes COPD medication and medical records will provide all that information. If medical records couldn't' be provided, CRC can collect this information by patients' recall.

- \* This will be evaluated by Clinical research coordinator (CRC) from the photo of the physicians' prescription collected from the patients.
- † Patient questionnaire is General self-efficacy scale. Patient's survey is developed by the study initiator Note: During the 3-month period, there might be changes in prescription, but only the current treatment prescribed to the patient and the patient's use of the treatment on the day or before the day of the call will be documented.

If the patient cannot be contacted telephonically at the first attempt, a minimum of 3 attempts should be made. This should be documented in a medical note. If the subject meets the conditions to withdraw from the project, no further data will be collected from the subject.

#### 3.2.2.2 Patients presenting with a moderate exacerbation (non-hospitalized)

## Baseline visit (Day 1)

Data will be collected as per stable patient in section 3.2.2.1- Baseline visit. If a  $FEV_1$  measurement from the last 6 months is not available, spirometry will be performed at the discretion of treating physician, dependent on whether it is possible or reasonable for the patient to do this.

#### 1-week follow-up (Day 8 ± 3)

This follow-up visit will be telephonic on day 8 (+3 days window). The patient will be interviewed to obtain the following details;

- 1. Any visit to hospital for COPD treatment in the last week? (Yes/No)
  - a. If Yes name of the hospital(s), physician's name, date(s) and physician
    prescription(s). These can be all collected by taking a picture of the prescription
- 2. CAT
- 3. Collect spontaneous AE/SAE reports on GSK products

If the patient cannot be contacted at first attempt, a minimum of 3 attempts should be made. This should be documented in a medical note.

## 3-month Follow-up (Day 90 ± 7)

Patients will be followed-up telephonically after 3 months. Data will be collected as per section 3.2.2.1- Follow-up visit for stable COPD patients.

Note: During the 3-month period, there might be changes in prescription, but only the current treatment prescribed to the patient and the patient's use of the treatment on the day or before the day of the call will be documented. If the subject meets the conditions to withdraw from the project, no further data will be collected from the subject.

#### 3.2.2.3 Patients requiring hospitalisation for an exacerbation

# Baseline visit (Day 1)

Baseline information as per section 3.2.2.1 will be collected on admission to the hospital, but if the patient is too ill, then baseline data will be collected before discharge. In the event that no historical  $FEV_1$  data within 6 months are available, spirometry will be performed if it is possible or reasonable for the patient to do. Dyspnoea, Eosinopenia, Consolidation, Acidaemia and atrial Fibrillation (DECAF) Score will be collected for the hospitalized patients during hospitalization period.

## Discharge Follow-up (Discharge day ± 1)

At the day of discharge (±1 day) patient will be interviewed face to face for obtaining data as follow;

- 1. Discharge date
- 2. COPD prescription at discharge (including the drugs prescribed this time and the drugs that the subject needs to continue to use)
- 3. CAT
- 4. Concomitant medication review
- 5. Total direct cost of the hospitalization
- 6. Medical insurance reimbursement amount
- 7. All other data under 3.2.2.1 (if not already collected)
- 8. Collect spontaneous AE/SAE reports on GSK products
- 9. Spirometry if no spirometry record within 6 months before baseline

## 3-month Follow-up (Day $90 \pm 7$ )

Patients will be followed-up telephonically after 3 months. Data will be collected as per section 3.2.2.1- Follow-up visit.

Note: During the 3-month period, there might be changes in prescription, but only the current treatment prescribed to the patient and the patient's use of the treatment on the day or the day before of the call will be documented. If the subject meets the conditions to withdraw from the project, no further data will be collected from the subject.

The sampling plans specified in sections 3.2.2.1-3.2.2.3 are summarised in Table 1.

Table 1: Visit & Observations recording

| Patients | Baseline Visit | 1-week Follow-up | 3-month |
|----------------|----------------|-------------------|----------------------|
| classification | | or discharge | Follow-up |
| | | Follow-up ±3 days | (Telephonic) ±7 days |

| Stable patients (Newly and previously diagnosed) Exacerbation Patients (Non-Admitted) | Demography, time since first COPD diagnosis, comorbidities, COPD exacerbation and medication history, concomitant medication, FEV1%pred, CAT score and mMRC, medicines prescribed at visit, smoking status, socio economic status, patient survey and questionnaire, physician survey, inhaler availability, spontaneous AE/SAE report collection, Maintenance treatment class availability in hospital internal pharmacy, prescribing physician's name. Demography, time since first COPD diagnosis, comorbidities, COPD exacerbation and medication history, concomitant medication, FEV1%pred*, CAT score and mMRC, medicines prescribed at visit, smoking status, socio economic status, patient survey and questionnaire, physician survey, inhaler availability, spontaneous AE/SAE report collection, Maintenance treatment class availability in hospital internal pharmacy, prescribing physician's name. | Telephone CAT score, any visit to hospital(Y/N), If Yes - name of the hospital(s), date(s) and physician prescription(s); spontaneous AE/SAE report collection | Telephone CAT score; current treatment taken by patient, the prescription of current treatment and time of prescription (or last hospital visit time and prescription); Name of hospital and name of physician; COPD clinic revisit times and reason, Frequency of COPD exacerbation between baseline visit and 3 months follow up, patient survey, concomitant medication review, spontaneous AE/SAE report collection |
|---|---|---|---|
| Exacerbation patients (Hospitalized)** | Demography, time since first COPD diagnosis, co- morbidities, COPD exacerbation and medication history, concomitant medication, FEV1%pred*, CAT score and mMRC, medicines | Onsite CAT score Prescription at discharge, discharge date spontaneous | |

| prescribed at visit, smoking status, socio economic status, Dyspnoea, Eosinopenia, Consolidation, Acidaemia and atrial Fibrillation (DECAF) Score, patient survey and questionnaire, physician survey, inhaler availability**, spontaneous AE/SAE report collection, Maintenance treatment class availability in hospital internal pharmacy, prescribing physician's name. | AE/SAE report collection, Concomitant medication, Total direct cost of the hospitalization, Medical insurance reimbursement amount |
|---|---|
|---|---|

<sup>\*</sup> If FEV1 data is not available, it will be performed at the discretion of treating physician/collected during discharge

#### 3.3 Data Source / Data Collection

## 3.3.1 Endpoints data source

# 3.3.1.1 Primary Endpoints

- The data source will be the study case record form (CRF)
- The prescription for COPD maintenance therapy, grouped into one or more of the
  following treatment classes: (Long-Acting Muscarinic Antagonist [LAMA], Long-Acting
  Beta-Agonist [LABA], dual bronchodilator, inhaled corticosteroid [ICS]/ Long-Acting BetaAgonist [LABA], triple therapy, theophylline and n-acetyl cysteine/carbocysteine) at
  baseline. The categories will be binary, e.g. treatment class used: Yes/No.
- COPD prescription for maintenance therapy collected at 3 months (all patients) and at 1 week after a moderate exacerbation or on discharge following hospitalisation.

## 3.3.1.2 Secondary Endpoints

- This will include the prescribing data listed in 3.3.1.1
- FEV1, exacerbations in previous 1 year, medication history within 1 month before baseline visit, CAT score, mMRC score, DECAF score in hospitalised patients, comorbidity, socio-economic status.
- The change in treatment over 3 months, (baseline medication will be used, as described, coupled with current prescribing collected at telephone interview at 3 months).

<sup>\*\*</sup> The baseline information can be collected at discharge



#### 3.3.2 Exposure and outcomes

#### 3.3.2.1 Demographics

- Sex: Male, Female
- Age, years (below 65 years old vs. 65 years old and above)
- Height, meters
- Weight, kg
- Body mass index (BMI=kg/m², BMI<18.5 underweight, BMI18.5~23.9 normal, BMI≥24 overweight, BMI≥28 obesity)</li>
- Smoking status: never a smoker; former smoker (previously smoked and has not smoked for at least 6 months prior to this visit); current smoker (10 pack years and smoked within 6 months of this visit); the number of pack years for former smoker and current smoker should be calculated (round up to the nearest integer)
- Co-morbid diseases: Cardiovascular Disease (CVD defined as ischemic heart disease, heart failure, atrial fibrillation, hypertension), Diabetes, Hyperlipemia, Anxiety, Depression, Gastroesophageal reflux disease (GERD), obstructive sleep apnea syndrome (OSAS), concurrent asthma with COPD, past history of tuberculosis.
- Class of maintenance treatment available at hospital internal pharmacy

# 3.3.2.2 COPD assessment test (CAT):

The CAT is an 8-item unidimensional measure of health status impairment in patients with COPD. It is applicable worldwide. The development of the CAT has involved well accepted methodologies used to develop psychometric tools [Jones, 2009a; Jones, 2009b]. With CAT, patients are scored on eight items (cough, phlegm, chest tightness, breathlessness, activity limitation, confidence, sleep and energy) on a scale of 0-5 depending on their impact. The sum of scores for each item gives the patient's impact score ranging from 0 [CCI

After being instructed how to use the CAT (following the COPD assessment test manual www.CATestonline.org), the subjects will complete it by themselves, without supervision or assistance from investigator. If the CAT is normally used by the investigator in their routine clinical work, they should use it as they would do normally; if the investigator does not

routinely use the CAT, it should be completed after the treatment decision has been made. The investigator should check whether the subjects complete all items before the patient leaves.

# 3.3.2.3 Modified British Medical Research Council (mMRC) Questionnaire

The mMRC was developed in 1960 [Fletcher, 1960], and relates well to other measures of health status [Bestall, 1999] and predicts future mortality risk [Sundh, 2012; Nishimura, 2002]. With mMRC, patients are scored on a scale of 0-4 depending on their disability due to shortness of breath from 0 ccl to 4 ccl

The mMRC will be completed by each patient by themselves, without supervision, after the CAT. If the mMRC is normally used by the investigator in their routine clinical work, they should use it as they would do normally; if the investigator does not routinely use the mMRC, it should be completed after the treatment decision has been made. The investigator should check whether the patient has completed the mMRC adequately but cannot assist in completing it.

## 3.3.2.4 Spirometry:

Spirometry data will be obtained for all patients at each site. If lung function data are available within the previous 6 months, this should be recorded, and no test will be required at the study visit. If previous FEV<sub>1</sub> data are not available and the patient cannot perform adequate spirometry because they are being hospitalized for an exacerbation, this will be performed before discharge from hospital.

Subjects should wear a nose clip while performing spirometry maneuvers. For  $FEV_1$  and FVC determinations, at least 3 acceptable spirometry efforts (with no more than 8) should be obtained. Acceptable spirometry efforts should have a satisfactory start of test and end of test (i.e, a plateau in the volume-time curve) and should be free from artifacts due to cough, early termination, poor effort, obstructed mouthpiece, equipment malfunction, or other reasons [

Miller, 2005; Pelligrino, 2005]. The largest FEV<sub>1</sub> and FVC from the 3 acceptable efforts should be recorded, even if they do not come from the same effort.

Based on the spirometry results, subjects will be stratified into airflow limitation category (Gold 1 - Gold 4) as per Table 2.

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

#### 3.3.2.5 Physician survey

Physician will be asked questions on why they follow their prescription practices. The survey will give brief idea on grounds which physicians prescribe treatment to patients.

- In addition to the severity of the patient's disease, which factors have influenced your prescription for THIS patient? (choose one or more options)
  - A. Patient or family 's economic condition
  - B. Patient's reimbursement position
  - C. Drug availability of your hospital
  - D. Patient's ability to use the inhaler
  - E. Patient's preference
- ➤ If none of the above factors applies, which treatment would you choose for THIS patient? (Choose one option)
  - A. None
  - B. SABA or SAMA (or both)
  - C. LAMA or LABA
  - D. LAMA+LABA
  - E. ICS+LABA
  - F. ICS+LABA+LAMA

## 3.3.2.6 Patient survey and questionnaire

To gain a better understanding of patient-related factors including socioeconomic status, knowledge of COPD and ideas on COPD treatment, a patient survey developed by the study initiator will be administered, together with questionnaires at the baseline visit and at the 3-month visit. The questionnaires will be administered in validated Chinese versions. These are physical activity, assessed using the International Physical Activity Questionnaire (IPAQ), mood state measured with the Patient Health Questionnaire (PHQ9), and self-efficacy using the, General Self-Efficacy Scale (see appendix for full details). The survey and questionnaires will deepen our understanding of the patients' behaviors and beliefs and how they influence adherence to treatment.

## 3.3.2.7 Exacerbation history and hospitalization for exacerbation in preceding year:

The patient's exacerbation history in the preceding year will be recorded. COPD exacerbation is an acute event characterized by a worsening of the patient's respiratory symptoms that is beyond normal day-to-day variations and leads to a change in medication [GOLD, 2019]. The

standard definition used in clinical studies requires a worsening of respiratory symptoms (including increased cough, sputum, breathlessness, chest tightness or wheeze) for 2 or more days.

The severity of the exacerbation will be determined using the following standard categories:

- 1. Mild a worsening of symptoms treated by the patient through an increase in use of their usual medicine, typically increased SABA use
- Moderate worsening of symptoms for which a patient seeks medical care and is treated by antibiotics and/or systemic corticosteroids/or corticosteroids nebulization
- 3. Severe –exacerbation requiring hospital admission.

#### 3.3.2.8 Safety

The data on AE/SAE should not be collected directly by physician. If an AE (serious or non-serious) or complaint with any specifically named GSK product is reported spontaneously by a patient during the course of the study, this will be documented by the site staff.

#### **3.3.2.9** Physician prescription-COPD-Related Medication

This will be collected by treatment class: Long-Acting Muscarinic Antagonist [LAMA], Long-Acting Beta-Agonist [LABA], dual bronchodilator, inhaled corticosteroid [ICS]/ Long-Acting Beta-Agonist [LABA], triple therapy, theophylline and n-acetyl cysteine/carbocysteine. Information which includes such COPD medication and related medical records will be request.

#### 3.3.2.10 Socioeconomic status

The objective questions will be asked to patients understand their socioeconomic status

- Education (illiteracy, primary school, junior mid-school, high-school, university)
- Living area (in city, outside city)
- Marriage condition
- Family total income in the past 12 months
- Individual total income in the past 12 months
- Economic support from others in the past 12 months
- Total health expenditure in the past 12 months
- Out-of-pocket health expenditure in the past 12 months
- COPD expenditure in the past 12 months
- Out-of-pocket COPD expenditure in the past 12 months
- National basic medical insurance
- Commercial insurance

#### **3.3.2.11 DECAF** score

The is a 5-point scale that uses items from the MRC dyspnoea scale, together with blood eosinophils ( $<0.05 \times 10^9$ /L, consolidation (pneumonia) on CXR, moderate or severe acidaemia (pH < 7.3) and presence or history of atrial fibrillation. It has been extensively tested and validated [Echevarria, 2016].

## 4 SAMPLE SIZE / POWER CALCULATIONS

The primary objective of the study is to understand the prescription pattern of COPD maintenance treatment in Tier 2 and Tier 3 hospitals in China. Around 1500 patients with COPD will be enrolled which includes stable patients and patients with COPD exacerbations (moderate and severe). All enrolled patients will be included in the analysis. This sample size was chosen to ensure adequate patient representation and provide sufficient size for reliable analysis of different patient groups and key subgroups.

It is estimated that 750 patients each from tier 2 and tier 3 hospitals will be enrolled to provide adequate representation on healthcare status for COPD in China. The target number of patients in each tier of hospital and patient groups is shown in Table 3. After 500 patients have been recruited, the numbers will be reviewed to assess whether adequate number of participants have been enrolled for patient in stable state or with COPD exacerbations in each tier of hospital. At this point, recruitment policy might be changed to ensure an adequate distribution of patients. Thereafter, recruitment to different patient groups will be monitored monthly and further corrective action taken if needed.

Table 3: Patient recruitment strategy (estimated distribution ratio)

| Patient group | Tier 2 hospital (% of total patients) | Tier 3 hospital (% of total patients) |
|---|---|---|
| Stable | 25% | 25% |
| Moderate acute or | 25% | 25% |
| Hospitalized exacerbation | | |

The secondary objective of this study is to examine factors (include baseline disease severity and baseline socio-economic factors) that are associated with different patterns of maintenance treatment. In the secondary analysis, we attempt to find significant association between disease severity (GOLD Group: A&B vs. C&D) and triple therapy at baseline for COPD patients.

Based on a previous study [Brusselle, 2015], about 24% COPD patients in Group A&B were prescribed triple therapy at diagnosis and about 46% COPD patients in Group C&D were prescribed triple therapy at diagnosis. The proportion of patients in Group A&B accounted for

66% of the total. We will use logistic regression to test this association and the parameters mentioned will be used for power calculation.

With a two-sided 5% level of significance and a sample size of 375subjects of each patient group in each Tier of hospital, we will have a power bigger than 98% for demonstrating a statistically significant result for the association between disease severity (GOLD Group: A&B vs. C&D) and triple therapy at baseline for COPD patients.

# 4.1 Hypotheses

The null hypothesis used to test the association between disease severity and triple therapy will be:

H0: There is no association between disease severity (GOLD grade: A&B vs. C&D) and triple therapy at diagnosis for COPD patients.

The alternative hypothesis will be:

H1: There is association between disease severity (GOLD grade: A&B vs. C&D) and triple therapy at diagnosis for COPD patients.

#### 5 DATA ANALYSIS CONSIDERATIONS

This section summarizes the statistical approaches that will be implemented to assess the study objectives. The descriptive statistical results will be displayed for Tier 2 and 3 hospitals separately for all the analyses. All analyses will be conducted using SAS, version 9.4 or above.

#### 5.1 Primary analyses

The primary objective of this study is to quantify the pattern of maintenance treatment prescribing in different patient groups in Tier 2 and 3 hospitals in China. Firstly, the number and percentage of patients who use the maintenance treatment at each visit will be summarized. Moreover, for those who use maintenance treatment, the number and percentage of patients will be summarized for each of the following pattern of maintenance treatment:

- Long-Acting Muscarinic Antagonist [LAMA]
- Long-Acting Beta-Agonist [LABA]
- Dual bronchodilator
- Inhaled corticosteroid [ICS]/ Long-Acting Beta-Agonist [LABA]
- Triple therapy
- Theophylline
- N-acetyl cysteine/carbocysteine

The results for patients with stable disease and patients with exacerbation at baseline will be analysed separately for the following visits: baseline visit, 1-week follow up (for moderate exacerbations) and discharge follow-up (for hospitalised exacerbations). The results for patients with stable disease and patients with exacerbation will be pooled together for analysis for 3-month follow-up visit. The percentage will be compared between stable and exacerbating patients by maintenance treatment.

## 5.2 Secondary analyses

The secondary objective of this study is to examine factors (include baseline disease severity and baseline socio-economic factors) that are associated with different patterns of maintenance treatment at baseline. Separate analyses will be performed for stable and exacerbating patients, since it is possible that the factors that influence a physician's choice of treatment may differ between the two conditions.

This part of analysis will be conducted in the group of the patients with stable disease and patients with exacerbation. The number and percentage of patients in each pattern of maintenance treatment will be summarized by the following factors:

- Age
- Gender: female/male
- Smoking history
- Any comorbidity
- Baseline GOLD 2019 grade: A/B/C/D
- Annual income
- Proportion of outpatient medical insurance
- Place of residence (in city, outside city)
- Educational level (illiterate, primary school, junior mid-school, high-school, university)
- Baseline FEV1 stage: I-IV

Multivariate logistic regression will be used to identify adjusted odds ratios (ORs) and 95% confidence intervals (95% CIs) for having a certain maintenance treatment versus none, using the above factors as covariates.

Another secondary objective is to assess the proportion of patients whose prescribed maintenance treatment was stepped up, stepped down, stopped, switched or remained the same across the different study time points. The number and percentage of patients whose prescribed maintenance treatment was stepped up, stepped down, stopped, switched or remained the same will be summarized for each visit.

The results for patients with stable disease and patients with exacerbation will be analysed separately. For those with exacerbation, the results for patients with a moderate exacerbation and patients requiring hospitalisation for an exacerbation will be further analysed separately.

The proportion of who have changed from one pattern of maintenance treatment at baseline to another pattern at 3-month will be summarized separately for the group of patients with stable disease at baseline and those with an exacerbation.

One more secondary objective is to assess the disease burden of the patients. The number and percentage of patients in different mMRC score intervals, CAT score intervals, numbers of historic exacerbation will be summarized according to the usage of different historic treatments. Moreover, mMRC score, CAT score and number of historic exacerbations will be summarized by mean and standard deviation in different patterns of maintenance treatment.

Another secondary objective is to assess the proportion of patients actually receiving each treatment class at 3 months.



#### 5.4 Other analysis

Safety information will be summarized.

#### **6** LIMITATIONS

- At least one site in each of the main province of China will be selected. However, only
  1-2 sites per province will be selected and these may not be fully representative of all
  the Tier 2 and 3 hospitals in each province.
- The study includes only those Tier 2 hospitals which at a minimum to have LAMA and ICS/LABA and spirometry available; however, this will not fully reflect COPD management in all Tier 2 hospitals, because not all currently have such drugs available.
- It is a 3-month follow-up study and the duration is adequate to measure short-medium term changes, but COPD requires lifelong treatment, so this reflects only a short period of a patient's management
- The adherence data is reliant on the patients accurate reporting of which prescribed treatments they are taking, there can be an underestimation or overestimation of adherence to medication.

#### 7 STUDY CONDUCT, MANAGEMENT & ETHICS

# 7.1 Ethics Committee/IRB Approval

This study will be conducted in accordance with GCP and all applicable regulatory requirements, including, where applicable, the current version of the Declaration of Helsinki.

The investigator is responsible for ensuring that this protocol, the site's informed consent form, and any other information that will be presented to potential subjects (e.g., advertisements or information that supports or supplements the informed consent) are reviewed and approved by the appropriate Independent Ethics Committee (IEC). The investigator agrees to allow the IEC direct access to all relevant documents. The IEC must be constituted in accordance with all applicable regulatory requirements. GSK will provide the investigator with relevant document(s)/data that are needed for IEC review and approval of the study. Before CRFs can be shipped to the site, GSK must receive copies of the IEC approval, the approved informed consent form, and any other information that the IEC has approved for presentation to potential subjects.

#### 7.2 Informed Consent

- The investigator or his/her representative will explain the nature of the study to the
  participant or his/her legally authorized representative and answer all questions
  regarding the study.
- Participants will be informed that their participation is voluntary. Participants or their legally authorized representative will be required to sign a statement of informed consent that meets the requirements of 21 CFR 50, local regulations, ICH guidelines,

Health Insurance Portability and Accountability Act (HIPAA) requirements, where applicable, and the IRB/IEC or study centre.

- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- A copy of the ICF(s) must be provided to the participant or the participant's legally authorized representative.

#### 7.3 Data Protection

Subject to participant consent, it is expected that patient number, date of birth, postal code and sex will be the only patient identifiable data that will be included in this transfer.

The data will be housed within secure servers. Access to information is restricted by role and is project specific. Data are analysed on these secure servers, and only the output may be extracted.

The output from this study will not include any individually identifiable data.

## 7.4 Personally Identifiable Information (PII)

All efforts will be made to ensure compliance with all applicable human subject protection and data protection laws in China and regulations in effect. To this end, all analytical datasets will be in a format that does not allow subjects to be identified, whether directly or through identifiers linked to the subject.

#### 7.5 Adverse Event (AE), Pregnancy Exposure, and Incident Reporting

If an AE (serious or non-serious) or complaint with any specifically with GSK product is reported spontaneously by a subject during the course of the study, the PI or site staff must report to GSK local safety department within 24 hours of first becoming aware of the event in accordance with SOP\_54834 Management of Adverse Event, Pregnancy Exposure, and Incident Reports from Human Subject Research.

Per SOP 52214 (Pharmacovigilance Planning for Epidemiology and Health Outcomes human subject research), a Pharmacovigilance Plan (PVP) is required for research with and without safety-related objectives.

#### 7.6 Legal Basis for Processing Individual Human Data

The authors confirm that study data is Individual Human Data (IHD) owned by GSK and that:

The proposed use of the IHD is **Study Use\*** as outlined in the patient consent.

\* Study Use means - the use of IHD is as stated in the original study protocol and/or aligned with the informed consent form to answer the study objectives and satisfy regulatory requirements and learn more about the product studied and the disease/condition studied. This includes bringing the product to market or maintaining market access, which includes working with government agencies, insurers or health care payers and aiding GSK's understanding of clinical efficacy, safety, or effectiveness of the product.

#### 8 PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

## **8.1** Target Audience

GSK stakeholders will require the information generated by this study, as well as contribute to the published literature. The results will be disseminated externally via manuscripts or presentations.

## 8.2 Study reporting and publications

Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the clinical study report. The investigator will be provided reasonable access to statistical tables, figures, and relevant reports and will have the opportunity to review the complete study results at a GSK site or other mutually agreeable location.

GSK will also provide the investigator with the full summary of the study results. The investigator is encouraged to share the summary results with the study subjects, as appropriate.

The results summary will be posted to the Clinical Study Register no later than 12 months after the last subject's last visit (LSLV) or sooner if required by legal agreement, local law or regulation. In addition, a manuscript will be submitted to a peer-reviewed journal for publication within 18 months of LSLV. When manuscript publication in a peer- reviewed journal is not feasible, further study information will be posted to the GSK Clinical Study Register to supplement the results summary.

A manuscript will be progressed for publication in the scientific literature if the results provide important scientific or medical knowledge.

#### 9 REFERENCES

Agusti AG. COPD, a multicomponent disease: implications for management. Respir Med. 2005 Jun;99(6):670-82.

Bestall JC, Paul EA, Garrold R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax 1999;54(7):581-6.

Brusselle, G, Price D, Gruffydd-Jones K, Miravittles M, Kleiner DL, Stewart R, et al. The inevitable drift to triple therapy in COPD: an analysis of prescribing pathways in the UK. International Journal of COPD. 2015; 10: 2207-2217

Cai S, Qin L, Tanoue L, Hu A, Jia X, Luo H, et al. Effects of one-hour training course and spirometry on the ability of physicians to diagnose and treat chronic obstructive pulmonary disease. PLoS One. 2015 Feb 23;10(2):e0117348.

COPD assessment test 2018, <a href="https://www.catestonline.org/">https://www.catestonline.org/</a>. Owned by GlaxoSmithKline

Davis JR, Wu B, Kern DM, Tunceli O, Fox KM, Horton J, et al. Impact of Nonadherence to Inhaled Corticosteroid/LABA Therapy on COPD Exacerbation Rates and Healthcare Costs in a Commercially Insured US Population. Am Health Drug Benefits. 2017 Apr;10(2):92-102.

Echevarria C, Steer J, Heslop-Marshall K, et al. Validation of the DECAF score to predict hospital mortality in acute exacerbations of COPD. Thorax 2016;71:133–40

Fang X, Li S, Gao L, Zhao N, Wang X, Bai C A short-term educational program improved physicians' adherence to guidelines for COPD and asthma in Shanghai. Clin Transl Med. 2012 Jul 3;1(1):13.

Fletcher CM. Standardised questionnaire on respiratory symptoms: a statement prepared and approved by the MRC committee on the Aetiology of Chronic Bronchitis (MRC breathless score). BMJ 1960;2:1662.

Global initiative for chronic obstructive lung disease (GOLDa). Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease (2019 report)

Global initiative for chronic obstructive lung disease (GOLD). Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease (2020 report)

Jia GH, Lu M, Wu R, Chen Y, Yao WZ. Gender difference on the knowledge, attitude, and practice of COPD diagnosis and treatment: a national, multicenter, cross-sectional survey in China. Int J COPD 2018; 13: 3269-3280

Jiangna H, Lu D, Nanshan Z, David Y. Breathlessness or Health Status in Chronic Obstructive Pulmonary Disease: The Impact of Different Definitions. COPD 2015, 12:115–125

Jones P, Harding G, Wiklund I, Berry P, Leidy N. Improving the process and outcome of care in COPD: development of a standardised assessment tool. Primary Care Resp J.2009 b; 18:208-215.

Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009a;34:648-654.

Li M, Wang F, Chen R, Liang Z, Zhou Y, Yang Y, et al. Factors contributing to hospitalization costs for patients with COPD in China: a retrospective analysis of medical record data. Int J Chron Obstruct Pulmon Dis. 2018 Oct 12;13:3349-3357.

Mäkelä MJ, Backer V, Hedegaard M, Larsson K. Adherence to inhaled therapies, health outcomes and costs in patients with asthma and COPD. Respir Med. 2013 Oct;107(10):1481-90.

Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J.Standardisation of spirometry. Eur Respir J, 2005;26:319-338.

Nishimura K, Oga T, Tsukino M, Hajiro T, Ikeda A, Jones PW. Reanalysis of the Japanese experience using the combined COPD assessment of the 2011 GOLD classification. Respiratory Investigation 2014;52:129-135.

Pelligrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R et al. Interpretative strategies for lung function tests. Eur Respir J. 2005;26:948-968.

Qaseem A, Wilt TJ, Weinberger SE, Hanania NA, Criner G, van der Molen T, et al. Diagnosis and management of stable chronic obstructive pulmonary disease: a clinical practice guideline update from the American College of Physicians, American College of Chest Physicians, American Thoracic Society, and European Respiratory Society. Ann Intern Med. 2011 Aug 2;155(3):179-91.

Restrepo RD, Alvarez MT, Wittnebel LD, Sorenson H, Wettstein R, Vines DL, et al. Medication adherence issues in patients treated for COPD. Int J Chron Obstruct Pulmon Dis. 2008;3(3):371-84

Rodríguez LA1, Wallander MA, Martín-Merino E, Johansson S. Heart failure, myocardial infarction, lung cancer and death in COPD patients: a UK primary care study. Respir Med. 2010 Nov;104(11):1691-9.
Rui T, Bian Y, Balwinder S, Liu Z, Wang T, Li G. Under diagnosis of COPD in high risk population in China American Journal of Respiratory and Critical Care Medicine 2014 189 (Meeting Abstracts)

Sundh J, Janson C, Lisspers K, Stallberg B, Montgomery S. The dyspnoea, Obstruction, Smoking, Exacerbation (DOSE) index is predictive of mortality in COPD. Prim Care Respir J 2012;21(3):295-301.

Toy EL, Beaulieu NU, McHale JM, Welland TR, Plauschinat CA, Swensen A, et al. Treatment of COPD: relationships between daily dosing frequency, adherence, resource use, and costs. Respir Med. 2011 Mar;105(3):435-41.

Wang C, Xu J, Yang L, Xu Y, Zhang X, Bai C, et al. Prevalence and risk factors of chronic obstructive pulmonary disease in China (the China Pulmonary Health [CPH] study): a national cross-sectional study. Lancet. 2018 Apr 28;391(10131):1706-1717.

Watz H, Tetzlaff K, Magnussen H, Mueller A, Rodriguez-Roisin R, Wouters EFM, Vogelmeier C, Calverley PMA. Spirometric changes during exacerbations of COPD: a post hoc analysis of the WISDOM trial. Respir Res. 2018 Dec 13;19(1):251.

Yang HY, Wu J, Zheng Y, Xie K, Jin L, Xie J, et al. Economic burden associated with acute exacerbations of chronic obstructive pulmonary disease in CHINA (abstract). Proceedings of the conference on, 'Value in health 15 (2012) A1 – A256

Zha Z, Leng R, Xu W, Bao H, Chen Y, Fang L, et al. Prevalence and risk factors of chronic obstructive pulmonary disease in Anhui Province, China: a population-based survey. BMC Pulm Med. 2019 May 29;19(1):102.

#### 10 APPENDICES

#### **10.1** Appendix 1: SCHEDULE OF ACTIVITIES

| Procedure | Baseli<br>ne<br>Visit | Dischar<br>ge<br>follow-<br>up for<br>admitte<br>d<br>patients | 1-week<br>follow up<br>for non-<br>admitted<br>patients<br>Day 8+3<br>(Telephon<br>e) | 3 months<br>follow up ±7<br>(Telephone) | Notes |
|---|---|---|---|---|---|
| Informed consent | Х | | | | |
| Inclusion and exclusion criteria | Х | | | | |
| Demography | Х | | | | |

| Full physical examination including height and weight | х | | | | |
|---|---|---|---|---|---|
| Co-morbidities | Х | | | | |
| COPD diagnosed history | Х | | | | |
| COPD exacerbation<br>history in prior 12<br>month | х | | | | |
| Current COPD disease condition (stable or acute) | х | | | | |
| Smoking history | Х | | | | |
| | | | | | a. will be collected |
| | | | | | from medical |
| | X | | | | records (will not be |
| District and the design | | | | | collected from |
| Physician name (code) | | | | | patients) |
| | | | | | a. COPD |
| | | | | | prescription when |
| | | | | | discharge<br>b. the latest COPD |
| | X | Xa | Xp | Xc | prescription at 1- |
| | ^ | X. | X | <b>X</b> | week follow up |
| | | | | | c. the latest COPD |
| | | | | | prescription at 3- |
| COPD prescription | | | | | month follow up |
| | | | | | a. within past 1 |
| Current COPD | Xa | | X | X | month before |
| medication | | | | | baseline visit |
| | | | | | a. will be collected |
| | | | | | from medical |
| | | | | | records or |
| | | | | Χa | patients' recall (the |
| Prescription date, | | | | | physician's name |
| physician and hospital | | | | | will not be |
| of current COPD | | | | | collected from |
| medication | | | | | patients) |
| | | | | | a. the lung function can be collected |
| Spirometry | Χ | Xa | | | before discharge if |
| | | | | | the patient's |

| | | | | | disease is too |
|---|---|---|---|---|---|
| | | | | | serious |
| DECAF score<br>assessment (admitted<br>patients) | X <sup>a</sup> | | | | a. can be assessed during hospitalization period |
| Physician's survey | X <sup>a</sup> | | | | a. to collect outpatients |
| Patient's survey and questionnaire | X | | | X | 1. Baseline period: Patient questionnaires include IPAQ, PHQ9, self-efficacy energy scale (GSE); baseline patient survey 2. 3-month follow- up period: patient questionnaires include self- efficacy energy scale (GSE); follow- up period patient survey |
| CAT | Х | Х | Х | Х | |
| mMRC Dyspnea Scale | Х | | | | |
| Socio-economic | Х | | | | |
| Insurance details | X | | | | |
| Inhaler availability | Х | | | | |
| Discharge time | | Х | | | |
| COPD Clinic revisit times and reason | | | Xa | Xa | a. If patient visits to clinic |
| Frequency of COPD exacerbation between baseline visit and 3 months follow up | | | | x | |
| Concomitant medication review | Х | Х | Х | X | |
| AE review | | X | | | *AE data will not<br>be collected<br>directly. A<br>physician can<br>document the<br>adverse event or |

| | | concern reported by the patients. |
|------------|---|-----------------------------------|
| | | *SAE data will not |
| | | be collected |
| | | directly. A |
| SAE review | X | physician can |
| SAL Teview | | document the |
| | | event or concern |
| | | reported by the |
| | | patients. |

| CCI - This section contained Clinical Outcome Asscopyright laws and therefore have been excluded. | sessment data collecti | on questionnaires or in | ndices, which are prote | ected by third party |
|---|---|---|---|---|

| CCI - This section contained Clinical Outcome As copyright laws and therefore have been excluded. | sessment data collection | questionnaires or indices, wh | nich are protected by third party |
|---|---|---|---|
| copyright laws and therefore have been excluded. | | | |

| CCI - This section contained Clinical Outc<br>and therefore have been excluded. | come Assessment data collection | questionnaires or indices, which ar | e protected by third party copyright laws |
|---|---|---|---|

| CCI - This section contained Clinic therefore have been excluded. | al Outcome Assessment da | ta collection questionnain | res or indices, which are pr | rotected by third party c | opyright laws and |
|---|---|---|---|---|---|

| CCI - This section contained Clinica<br>herefore have been excluded. | al Outcome Assessment dat | ta collection questionnaires | or indices, which are protect | ted by third party copyright law | vs and |
|---|---|---|---|---|---|

| CCI - This sec | tion contain | ed Clinical | Outcome A | ssessment c | lata collection | on question | naires or in | dices, which | ch are prote | ected by thire | d party copyri | ght laws and |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

| CCI - This section contained Clinical and therefore have been excluded. | Outcome Assessment data | a collection questionnaire | s or indices, which are prot | ected by third party copyright laws |
|---|---|---|---|---|

| CCI - This section contained Clinica<br>herefore have been excluded. | d Outcome Assessment data co | illection questionnaires or indic | ees, which are protected by third | party copyright laws and |
|---|---|---|---|---|

| CCI - This section contained Cl therefore have been excluded. | inical Outcome Assessmen | t data collection question | nnaires or indices, which | are protected by third pa | rty copyright laws and |
|---|---|---|---|---|---|

| CCI - This section contained Clir<br>therefore have been excluded. | nical Outcome Assessment d | ata collection questionnai | ires or indices, which are p | rotected by third party co | pyright laws and |
|---|---|---|---|---|---|

| CCI - This section contained Clini<br>therefore have been excluded. | ical Outcome Assessment | data collection questionna | aires or indices, which a | re protected by third pa | rty copyright laws and |
|---|---|---|---|---|---|

| CCI - This section contained Clinical on therefore have been excluded. | Outcome Assessment da | nta collection questions | naires or indices, which | are protected by third | party copyright laws |
|---|---|---|---|---|---|

| CCI - This section contained Clinical Outcome Assessment data collection quest: and therefore have been excluded. | ionnaires or indices, which are protected by | third party copyright laws |
|---|---|---|
| and therefore have been excluded. | | |

| CCI - This section contained Clinical Outcom<br>and therefore have been excluded. | e Assessment data collectio | n questionnaires or indices, | , which are protected by the | ird party copyright laws |
|---|---|---|---|---|

| CC<br>exc | CI - This section contained Cluded. | linical Outcome Assessment | t data collection question | maires or indices, which | are protected by third pa | rty copyright laws and | therefore have bee |
|---|---|---|---|---|---|---|---|



10.6 Appendix 6: sPVP and PVP APPROVAL FORM

## **Study-Specific Pharmacovigilance Plan (sPVP)**

| Unique Identifier | 213550 |
|---|---|
| Full title of protocol | COPD disease burden, patient characteristics, maintenance |
| | treatment patterns and factors influencing treatment decisions |
| | in China Tier 2 and Tier 3 hospitals |
| Abbreviated title of protocol | COPD maintenance treatment patterns in China |
| Department | China Medical Respiratory TA |
| Study Accountable Person | PPD |
| Type of Study | Interventional (interaction) study with data collection - |
| (tick type of study that | face-to-face or phone-based interviews |
| applies) | Interventional (interaction) study with data collection - |
| | digital or paper surveys |
| | Non-interventional study with data collection where data |
| | source includes identifiable patient information (e.g., data |
| | extraction from medical records, existing registry) |
| | Other, please describe: Low-interventional study with data |
| | collection where data source includes identifiable patient |
| | information (e.g., data extraction from medical records, existing |
| | registry) |
| Study-Specific | 24-Aug-2020 |
| Pharmacovigilance Plan | |
| Approval Date | |
| Safety and Medical | PPD |
| Governance (SMG) | |
| Representative: | |

## **Revision Chronology:**

| Version Date | Document Type | Change(s) since last version |
|------------------------------|---------------|------------------------------|
| Enter original sPVP approval | Original | n/a |
| date | | |
| Enter amended sPVP | NA | NA |
| approval date | | |

| t(tick applicable statements) N/A - No supplier/vendor involved that could identify Human Safety Information (HSI) following exposure of GSK/ViiV products Supplier PV training will be conducted using the agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. N/A - No Investigator and/or site staff involved that could be in receipt of Human Safety Information (HSI) following exposure of GSK/ViiV products N/A - No Investigator and/or site staff involved that could be in receipt of Human Safety Information (HSI) following exposure of GSK/ViiV products Investigator and/or site staff PV training will be conducted using the agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. SAP is responsible for the collection, reporting, and reconciliation process for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR | 5) (5.5) | Study-Specific Pharmacovigilance Plan (sPVP) |
|---|---|---|
| Supplier PV training Information (HSI) following exposure of GSK/ViIV products Supplier/vendor PV training will be conducted using the agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. N/A – No Investigator and/or site staff involved that could be in receipt of Human Safety Information (HSI) following exposure of GSK/ViIV products N/A – No Investigator and/or site staff PV training will be conducted using the agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. SAP is responsible for the collection, reporting, and reconciliation process for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR | sPVP Element | |
| Supplier/vendor PV training will be conducted using the agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. N/A – No Investigator and/or site staff involved that could be in receipt of Human Safety Information (HSI) following exposure of GSK/ViiV products Investigator and/or site staff PV training will be conducted using the agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. SAP is responsible for the collection, reporting, and reconciliation process for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR | | ☐ N/A – No supplier/vendor involved that could identify Human Safety |
| training and current, approved content, prior to beginning the study. Training will be completed annually and documented. N/A - No Investigator and/or site staff involved that could be in receipt of Human Safety Information (HSI) following exposure of GSK/ViiV products Investigator and/or site staff involved that could be in receipt of Human Safety Information (HSI) following exposure of GSK/ViiV products Investigator and/or site staff PV training will be conducted using the agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. SAP is responsible for the collection, reporting, and reconciliation process for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR | | Information (HSI) following exposure of GSK/ViiV products |
| and current, approved content, prior to beginning the study. Training will be completed annually and documented. N/A – No Investigator and/or site staff involved that could be in receipt of Human Safety Information (HSI) following exposure of GSK/ViiV products agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. SAP is responsible for the collection, reporting, and reconciliation process for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR HSI Collection Processes HSI Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of saset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | Supplier/vendor PV training will be conducted using the agreed method |
| N/A − No Investigator and/or site staff involved that could be in receipt of Human Safety Information (HSI) following exposure of GSK/ViiV products Investigator and/or site staff PV training will be conducted using the agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. SAP is responsible for the collection, reporting, and reconciliation process for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR | training | and current, approved content, prior to beginning the study. Training will be |
| Investigator and site staff PV training Human Safety Information (HSI) following exposure of GSK/ViiV products Investigator and/or site staff PV training will be conducted using the agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. SAP is responsible for the collection, reporting, and reconciliation process for HSI. | | completed annually and documented. |
| and site staff PV training Investigator and/or site staff PV training will be conducted using the agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. SAP is responsible for the collection, reporting, and reconciliation process for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR The protocol includes the rationale for collection of specific types of adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | N/A – No Investigator and/or site staff involved that could be in receipt of |
| PV training agreed method and current, approved content, prior to beginning the study. Training will be completed annually and documented. SAP is responsible for the collection, reporting, and reconciliation process for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR HSI Collection Processes The protocol includes the rationale for collection of specific types of adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | Investigator | Human Safety Information (HSI) following exposure of GSK/ViiV products |
| Training will be completed annually and documented. SAP is responsible for the collection, reporting, and reconciliation process for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR HSI Collection Processes HSI Reporting Processes Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | and site staff | ☐ Investigator and/or site staff PV training will be conducted using the |
| Safety- specific roles SAP is responsible for the collection, reporting, and reconciliation process for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR The protocol includes the rationale for collection of specific types of adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | PV training | agreed method and current, approved content, prior to beginning the study. |
| Safety- specific roles for HSI. Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR HSI Collection Processes HSI Reporting Processes OR The protocol includes the rationale for collection of specific types of adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | Training will be completed annually and documented. |
| specific roles Supplier/vendor is responsible for the collection, reporting, and reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product | | SAP is responsible for the collection, reporting, and reconciliation process |
| reconciliation process for HSI. The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR The protocol includes the rationale for collection of specific types of adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy SGSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | Safety- | for HSI. |
| Source The protocol includes details about collection of HSI, including all adverse reaction/event, following exposure to any GSK/ViiV product OR The protocol includes the rationale for collection of specific types of adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: | specific roles | Supplier/vendor is responsible for the collection, reporting, and |
| reaction/event, following exposure to any GSK/ViiV product OR HSI Collection Processes The protocol includes the rationale for collection of specific types of adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | reconciliation process for HSI. |
| HSI Collection Processes The protocol includes the rationale for collection of specific types of adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy OR GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | The protocol includes details about <b>collection</b> of HSI, including all adverse |
| HSI Collection Processes The protocol includes the rationale for collection of specific types of adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | reaction/event, following exposure to any GSK/ViiV product |
| HSI Collection Processes The protocol includes the rationale for collection of specific types of adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | |
| AE, pregnancy Adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy SGSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | OR |
| AE, pregnancy Adverse reaction/event (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy SGSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | |
| AE, pregnancy Required rescond option (e.g. objectives of the study, the stage of the asset development, level of clinical oversight). Required response if second option is selected: The rationale for the collection of data differs from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy SCSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | The protocol includes the rationale for <b>collection</b> of specific types of |
| development, level of clinical oversight). Required response if second option is selected: ☐ The rationale for the <b>collection</b> of data <u>differs</u> from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options ☐ The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR ☐ The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy ☐ GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | adverse reaction/event (e.g. objectives of the study, the stage of the asset |
| The rationale for the <b>collection</b> of data <u>differs</u> from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | Processes | development, level of clinical oversight). |
| The rationale for the <b>collection</b> of data <u>differs</u> from minimum criteria, this has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | |
| has been approved by the Central Safety Department. Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | Required response if second option is selected: |
| Please select one of the following options The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | The rationale for the <b>collection</b> of data <u>differs</u> from minimum criteria, this |
| The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy SK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | has been approved by the Central Safety Department. |
| The protocol includes details about reporting of all HSI following exposure of GSK/ViiV products. HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy SK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | |
| HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | Please select one of the following options |
| HSI Reporting Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | The protocol includes details about reporting of all HSI following exposure |
| Processes OR The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | of GSK/ViiV products. |
| The protocol includes details about the rationale for reporting (e.g., objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | HSI Reporting | |
| objectives of the study, the stage of asset development, level of clinical oversight) targeted follow-up requirements AE, pregnancy GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | Processes | OR |
| oversight) targeted follow-up requirements AE, pregnancy SSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | The protocol includes details about the rationale for reporting (e.g., |
| AE, pregnancy SSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting | | objectives of the study, the stage of asset development, level of clinical |
| | | oversight) targeted follow-up requirements |
| exposure, and Form for Epidemiology and Health Outcome studies | AE, pregnancy | GSK Global Adverse Event, Pregnancy Exposure, and Incident Reporting |
| | exposure, and | Form for Epidemiology and Health Outcome studies |

| sPVP Element | Study-Specific Pharmacovigilance Plan (sPVP) |
|---|---|
| SPVP LIEITIETIC | (tick applicable statements) |
| incident | Alternative collection form(s) will be utilized |
| collection | (if ticked, please specify the form title here - e.g. standard clinical trial SAE |
| forms | form, Pregnancy Notification Form, and/or any additional study/product- |
| | specific safety data collection form, if appropriate) |
| | ☐ N/A – No batch reviewing of the data. |
| | Batch review will be conducted |
| Frequency of | (if ticked, please specify the frequency of review) |
| data review | During the visit and follow-ups in this study, once AEs, pregnancy exposures |
| | is identified, the investigator will collect and report. |
| | Specify review and timing for the communication of study results to SMG |
| | For serious related AE (SADR) or pregnancy exposure safety report sent to |
| Reviewing | local PV team, the report would be forwarded to the global service provider |
| and reporting | (IQVIA) for their further processing to the drug safety headquarters (CSD) |
| study results | within 24 hours (the next working day in case of weekends); For non serious |
| | related AE (ADR), the report would be forwarded to the global service |
| | provider (IQVIA) for their further processing to the drug safety headquarters |
| | (CSD) within 5 calendar days. |
| | 1 ' ' |
| Interim study | N/A – No interim study reports are planned. |
| Interim study reports | <ul> <li>N/A − No interim study reports are planned.</li> <li>Interim study reports will be shared with the SERM product specialist /</li> </ul> |
| - | N/A – No interim study reports are planned. |
| - | <ul> <li>N/A − No interim study reports are planned.</li> <li>Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> </ul> |
| - | <ul> <li>N/A − No interim study reports are planned.</li> <li>Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>Reconciliation process defined in protocol</li> <li>Reconciliation process defined in sPVP, please describe</li> </ul> |
| reports | <ul> <li>N/A − No interim study reports are planned.</li> <li>Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>Reconciliation process defined in protocol</li> </ul> |
| reports | <ul> <li>N/A − No interim study reports are planned.</li> <li>Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>Reconciliation process defined in protocol</li> <li>Reconciliation process defined in sPVP, please describe</li> <li>Study manager is responsible for sending AE reconciliation form to local PV team monthly.</li> </ul> |
| reports | <ul> <li>N/A − No interim study reports are planned.</li> <li>Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>Reconciliation process defined in protocol</li> <li>Reconciliation process defined in sPVP, please describe</li> <li>Study manager is responsible for sending AE reconciliation form to local PV team monthly.</li> <li>Local PV team will assist in forwarding the AE reconciliation form to the</li> </ul> |
| Reconciliation process | <ul> <li>N/A − No interim study reports are planned.</li> <li>Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>Reconciliation process defined in protocol</li> <li>Reconciliation process defined in sPVP, please describe</li> <li>Study manager is responsible for sending AE reconciliation form to local PV team monthly.</li> <li>Local PV team will assist in forwarding the AE reconciliation form to the case management group (CMG), CMG is responsible for checking.</li> </ul> |
| Reconciliation process | <ul> <li>N/A − No interim study reports are planned.</li> <li>Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>Reconciliation process defined in protocol</li> <li>Reconciliation process defined in sPVP, please describe</li> <li>Study manager is responsible for sending AE reconciliation form to local PV team monthly.</li> <li>Local PV team will assist in forwarding the AE reconciliation form to the case management group (CMG), CMG is responsible for checking.</li> <li>SAP will review the sPVP elements and discuss during regular study team</li> </ul> |
| Reconciliation process PVP monitoring | <ul> <li>N/A − No interim study reports are planned.</li> <li>Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>Reconciliation process defined in protocol</li> <li>Reconciliation process defined in sPVP, please describe</li> <li>Study manager is responsible for sending AE reconciliation form to local PV team monthly.</li> <li>Local PV team will assist in forwarding the AE reconciliation form to the case management group (CMG), CMG is responsible for checking.</li> <li>SAP will review the sPVP elements and discuss during regular study team and/or supplier meetings to ensure the plan is working effectively.</li> </ul> |
| Reconciliation process | <ul> <li>N/A – No interim study reports are planned.</li> <li>☐ Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>☐ Reconciliation process defined in protocol</li> <li>☑ Reconciliation process defined in sPVP, please describe</li> <li>● Study manager is responsible for sending AE reconciliation form to local PV team monthly.</li> <li>● Local PV team will assist in forwarding the AE reconciliation form to the case management group (CMG), CMG is responsible for checking.</li> <li>☑ SAP will review the sPVP elements and discuss during regular study team and/or supplier meetings to ensure the plan is working effectively.</li> <li>☐ Other, please describe</li> </ul> |
| Reconciliation process PVP monitoring process | <ul> <li>N/A – No interim study reports are planned.</li> <li>☐ Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>☐ Reconciliation process defined in protocol</li> <li>☑ Reconciliation process defined in sPVP, please describe</li> <li>• Study manager is responsible for sending AE reconciliation form to local PV team monthly.</li> <li>• Local PV team will assist in forwarding the AE reconciliation form to the case management group (CMG), CMG is responsible for checking.</li> <li>☑ SAP will review the sPVP elements and discuss during regular study team and/or supplier meetings to ensure the plan is working effectively.</li> <li>☐ Other, please describe</li> <li>☐ Defined in protocol</li> </ul> |
| Reconciliation process PVP monitoring process Provision of | <ul> <li>N/A – No interim study reports are planned.</li> <li>☐ Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>☐ Reconciliation process defined in protocol</li> <li>☑ Reconciliation process defined in sPVP, please describe</li> <li>• Study manager is responsible for sending AE reconciliation form to local PV team monthly.</li> <li>• Local PV team will assist in forwarding the AE reconciliation form to the case management group (CMG), CMG is responsible for checking.</li> <li>☑ SAP will review the sPVP elements and discuss during regular study team and/or supplier meetings to ensure the plan is working effectively.</li> <li>☐ Other, please describe</li> <li>☐ Defined in protocol</li> <li>☑ Defined in sPVP, please describe</li> </ul> |
| Reconciliation process PVP monitoring process Provision of final study | <ul> <li>N/A – No interim study reports are planned.</li> <li>☐ Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>☐ Reconciliation process defined in protocol</li> <li>☐ Reconciliation process defined in sPVP, please describe</li> <li>• Study manager is responsible for sending AE reconciliation form to local PV team monthly.</li> <li>• Local PV team will assist in forwarding the AE reconciliation form to the case management group (CMG), CMG is responsible for checking.</li> <li>☐ SAP will review the sPVP elements and discuss during regular study team and/or supplier meetings to ensure the plan is working effectively.</li> <li>☐ Other, please describe</li> <li>☐ Defined in protocol</li> <li>☐ Defined in sPVP, please describe</li> <li>• All serious and non-serious AEs, pregnancy exposures, and incidents</li> </ul> |
| Reconciliation process PVP monitoring process Provision of | <ul> <li>N/A – No interim study reports are planned.</li> <li>☐ Interim study reports will be shared with the SERM product specialist / physician for review of the interim report safety data</li> <li>☐ Reconciliation process defined in protocol</li> <li>☑ Reconciliation process defined in sPVP, please describe</li> <li>• Study manager is responsible for sending AE reconciliation form to local PV team monthly.</li> <li>• Local PV team will assist in forwarding the AE reconciliation form to the case management group (CMG), CMG is responsible for checking.</li> <li>☑ SAP will review the sPVP elements and discuss during regular study team and/or supplier meetings to ensure the plan is working effectively.</li> <li>☐ Other, please describe</li> <li>☐ Defined in protocol</li> <li>☑ Defined in sPVP, please describe</li> </ul> |

# Study-specific Pharmacovigilance Plan (sPVP) Approval Page for: 213550

### **Approval**

I confirm that this sPVP is appropriate for the above study and has been completed in accordance with SOP 52214.

| Name | Job Title or Role & Qualification | Signature | Date |
|------|-----------------------------------|-----------|---------------|
| | | | (dd-mmm-yyyy) |
| | | | ļ |

Please forward this signed copy by e-mail to the Study Accountable Person and cc the sPVP mailbox: <u>Epi & HO PVP Queries@gsk.com</u>